CLINICAL TRIAL: NCT01776216
Title: Impact of Dairy Consumption on Hypertension: a Clinical Study.
Acronym: PLAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Patrick Couture, MD, FRCP, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: INAF-C11-02-163
Record Dates: First submitted 2013-01-21; First posted 2013-01-28 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Endothelial function; Dairy
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Dairy Products; Milk; Cheese

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dairy diet (Experimental): During the DAIRY diet, subjects will be asked to incorporate 3 servings of dairy into their everyday diet.
  Interventions: Other: Dairy diet
- Control diet (Placebo Comparator): During the CONTROL diet of the study, participants will be asked to consume energy equivalent replacement products into their everyday diet.
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Dairy diet — During the DAIRY diet, subjects will be asked to incorporate 3 servings of dairy: 375 ml of reduced fat milk (1% fat), 175 g of low fat yogurt (1.5% fat) and 30g of regular cheese (34% fat) into their every day diet.
  Other Names: Dairy products; Milk; Yogourt; Cheese
  Arms: Dairy diet
Other: Control diet — During the CONTROL diet of the study, participants will be asked to consume energy equivalent replacement products (290 ml of fruit juice, 156 ml of vegetable juice, 1 homemade cookie, 20g of cashew).
  Arms: Control diet

SUMMARY:
Hypertension and endothelial dysfunction are being increasingly recognized as key etiological factors in the development of atherosclerosis and subsequent cardiovascular disease (CVD). A substantial body of evidence indicates that treating patients with elevated blood pressure (BP) leads to marked reduction in the risk of stroke, myocardial infarction, heart failure, and renal failure. There is also accumulating evidence associating endothelial dysfunction, which is defined as incapacity of the arteries to vasodilate when required, to elevated BP and an increased risk of CVD.

While there are more and more studies on how diet affects BP in healthy subjects, the impact of dairy consumption per se on both endothelial function and ambulatory BP has not been well characterized in patients with established essential hypertension. Therefore, the general objective of the study is to investigate in a single-blind randomized controlled study the impact of dairy consumption on ambulatory BP and endothelial function in subjects with mild to moderate essential hypertension.

DETAILED DESCRIPTION:
The proposed research will be undertaken as a single-center randomized cross-over controlled study. A total of 80 men and women with mild to moderate essential hypertension but otherwise healthy will consume two 4-week diets, one rich in dairy and one without dairy, while consuming a diet low in saturated fat (<10% energy), in trans fat (<1% energy) and in cholesterol (<200 mg/day). During the DAIRY diet, subjects will be asked to incorporate 3 servings of dairy (milk, yogurt, cheese) into their every day diet. During the CONTROL arm of the study, participants will be asked to consume energy equivalent replacement products. The primary analysis consists in comparing mean daytime ambulatory BP values and endothelial function between the two treatments.

A 2-week stabilization run-in period will precede the randomization of participants. During this run-in period, participants will be asked and instructed to adapt their diet to a prudent dietary pattern low in saturated fat (<10% energy), in trans fat (<1% energy) and in cholesterol (<200 mg/day). The total amount of fat in the diet will not be restricted, with recommendations ranging from 25-35% of energy. However, substitution of saturated for unsaturated fat will be advocated. Sodium intake <2300 mg/d will also be recommended. Recommendations will also include advice on how to restrict the consumption of processed and energy dense foods. This 2-week run-in period will allow participants to familiarize themselves with the dietary recommendations used during the intervention per se. The two diets will be separated by a 4-week wash out period and will also consist to the prudent dietary pattern recommended. It must be stressed that foods will not be provided during the run-in and wash-out periods. These periods are imposed to minimize the inter- and intra-individual variability before and between the experimental phases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 70 years
* Mean daytime systolic blood pressure ≥ 135 mm Hg and ≤ 160 mm Hg
* Mean daytime diastolic blood pressure ≤ 110 mm Hg
* Consumption of dairy products fewer than 2 servings per day

Exclusion Criteria:

* Mean daytime systolic blood pressure > 160 mm Hg
* Mean daytime diastolic blood pressure > 110 mm Hg
* Dairy intake > 2 serving per day
* Smokers (>1 cigarette/day)
* Body weight variation >10% during the last 6 months prior to the study baseline
* BMI >35 kg/m2
* Previous history of cardiovascular disease, type 2 diabetes and monogenic dyslipidemia
* Subject taking anti-inflammatory drugs
* Subject with endocrine or gastrointestinal disorders
* Allergy, intolerance or aversion to dairy
* Clinical use of vitamin D or calcium supplements
* Vegetarians

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in mean daytime systolic blood pressure | At the fisrt visit of the study (screening) and at the end of the two 4-weeks diets (week 4 and week 12)
  Mean daytime systolic blood pressure will be measured by 24-h ambulatory blood pressure monitoring using the Spacelabs 90207 (Spacelabs, Inc., Redmond, WA)

SECONDARY OUTCOMES:
Change in mean daytime diastolic blood pressure | At the first visit of the study (screening) and at the end of the two 4-weeks diets (week 4 and week 12)
  Mean daytime diastolic blood pressure will be measured by 24-h ambulatory blood pressure monitoring using the Spacelabs 90207 (Spacelabs, Inc., Redmond, WA)
Change in endothelial function | At the end of the two 4-weeks diets (week 4 and week 12)
  Digital pulse amplitude will be measured with a PAT device placed on the tip of each index finger (Endo-PAT2000, Itamar Medical, Caesarea, Israel)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD,FRCP,PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutraceuticals and Functional Foods (INAF), Québec, Quebec, Canada

REFERENCES:
- [Derived] Drouin-Chartier JP, Gigleux I, Tremblay AJ, Poirier L, Lamarche B, Couture P. Impact of dairy consumption on essential hypertension: a clinical study. Nutr J. 2014 Aug 14;13:83. doi: 10.1186/1475-2891-13-83. PMID 25123170